CLINICAL TRIAL: NCT07082907
Title: Effects of Pet Therapy on Anxiety, Pulse Rate and Saturation In Children Between 3 and 6 Years of Age Who Received Nebulizer Treatment in the Emergency Department: A Randomized Controlled Study
Brief Title: Use Of Pet Therapy In Chıldren Receıvıng Nebulızer Treatment
Status: Completed | Type: Observational
Sponsor: Recep Tayyip Erdogan University (Other)
Responsible Party: Principal Investigator, Yağmur AKBAL DEMİRCİ, İnternal Medicine Nursing, Recep Tayyip Erdogan University
Other Study IDs: RTEU-SBF-YA-01
Record Dates: First submitted 2025-07-03; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-07

CONDITIONS: Respiratory Disease
Keywords: Respiratory disease; therapy animals; nebülizer; child
MeSH Terms: conditions — Respiration Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 3 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Control group: Control group; Standard application was provided to the children in the control group during the use of nebulizer. Fish in a bowl application was not given. However, in order to prevent bias in the study, children in the control group were also provided contact with fish after all data related to the study were collected.
  Interventions: Other: intervention group

INTERVENTIONS:
Other: intervention group — Before using the nebulizer, children were given 2 fish in a bowl accompanied by their parents. The child patient was in the fowler/semifowler position, the movements of the fish were monitored during the nebulization period, and the fish was fed by the child during this process (Communication was provided for at least 5 minutes.)

SUMMARY:
The use of nebulizers in children is one of the most common noninvasive methods used in respiratory system diseases. This application can cause anxiety and stress in children in hospital environments, especially in emergency departments. Our aim in this study is to evaluate the effect of pet therapy on anxiety, pulse and saturation in children between the ages of 3-6 who receive nebulizer treatment in units such as emergency departments.

DETAILED DESCRIPTION:
With nebulizer drug application, drugs such as bronchodilators, antibiotics, anticholinergics, corticosteroids are delivered directly to the lungs by inhalation. In nebulizer drug applications, the amount of drug, the method of administration, the duration, and the position of the patient are the most important criteria to be followed in order to administer the drug appropriately and effectively. Any disruption in any of these applications negatively affects the treatment process. Stress and anxiety experienced during nebulizer treatment in children can cause undesirable results in vital signs such as pulse. Treatment can therefore cause disruption. Although this application does not cause pain, being in a hospital environment and being an intervention applied by health professionals can cause anxiety in children. In addition, symptoms such as tachycardia are observed in children with some drugs administered via nebulizer. Many animal applications are used in animal-assisted therapies and it is emphasized that the stress of child patients decreases with these methods. In nebulizer drug use, the anxiety experienced by children due to both the mask and drug interactions applied in drug treatment and the changes in vital signs they encounter due to drug interactions have been tried to be supported with changing applications in the literature. However, when we look at the literature, we have not found any studies using pet therapy during nebulizer use.

ELIGIBILITY:
* Receiving inhalation therapy as an outpatient in the emergency department
* Between 3 and 6 years of age (determined as the age range in which children can communicate visually and emotionally)
* Parents must have received nebulizer training before the procedure/nurse-assisted treatment if this is the first procedure
* No visual impairment (for communication in pet therapy)
* No congenital cardiac disease (for homogeneous data in pulse and SpO2 monitoring)
* Agreeing to participate in the study

Exclusion criteria for the study:

* Children under 3 and over 6
* Parents and children who do not agree to participate in the study

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: This study will be conducted on 3-6 year old children who were admitted to a pediatric emergency unit of a training and research hospital with any respiratory distress and were recommended nebule therapy.
Sampling Method: Probability Sample
Enrollment: 60 (Actual)
Dates: Start 2025-02-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Scale for Assessing Children's Emotional Expression | The treatment period for the sick child in the emergency unit covers an average of 20-30 minutes during which time he/she receives nebulization.
  There was a significant relationship between the child's age and the annual number of nebulizer uses on the CDBDS scale score during Pet therapy application (R=0.547, R2=0.300, p<0.05).

OTHER OUTCOMES:
Scale for Assessing Children's Emotional Expression | Between February and June 2025
  The emergency department has varying levels of nebulization throughout the day. Some days, there are no patients at all, while other days, two or three pediatric patients receive nebulization. Reaching the sample size within this timeframe was among the other goals.

CONTACTS AND LOCATIONS:
Locations (1):
- Recep Tayyip Erdoğan University Training and Research Hospital, Rize, Centre, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Since this study is considered to be forward-looking, it is considered to be shared for now.